CLINICAL TRIAL: NCT02855385
Title: Health-seeking Behavior and Barriers to Care in Patients With Rectal Bleeding in Nigeria
Brief Title: Barriers to Care in Patients With Rectal Bleeding in Nigeria
Status: Completed | Type: Observational
Sponsor: Obafemi Awolowo University Teaching Hospital (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); University of Ilorin Teaching Hospital (Other); University College Hospital, Ibadan (Other)
Responsible Party: Principal Investigator, Olusegun Alatise, Consultant Surgeon/Senior Lecturer, Obafemi Awolowo University Teaching Hospital
Other Study IDs: ERC/2013/09/01
Record Dates: First submitted 2016-07-28; First posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Colorectal Cancer
Keywords: Rectal bleeding, , ,; Attitude; Health seeking behaviour; Nigeria; Screening; high risk patients
MeSH Terms: conditions — Colorectal Neoplasms; Gastrointestinal Hemorrhage; Behavior; Health Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patient group: This are patients who have current or previous history of rectal bleeding
- General Practitioner group: This are General practitioner who are in public or private hospitals who treat patients with rectal bleeding

SUMMARY:
This study sought to find the health seeking behavior of patients with rectal bleeding as related to their risk to develop colorectal cancer and also assess the general practitioner's perceived barriers to colonoscopy for patients with bleeding per rectum.

DETAILED DESCRIPTION:
Patients who had rectal bleeding are invited to electronic media and print media will be invited for free medical consultation. Consented patients will complete a purposely design questionnaire for the study to assess the knowledge, attitude and practice of patient with rectal bleeding as regard the possibility of occurrence of colorectal cancer.

General practitioners in three cities will be contacted to assess their screening strategy for patients with rectal bleeding

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with rectal bleeding that persisted for up to one month

Exclusion Criteria:

* Patient that has the cause of rectal bleeding already determined before presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with Rectal bleeding who consented to the study
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2013-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Knowledge score in relations to the demographics of patients with rectal bleeding | 60 days
  To investigates patients' knowledge of the causes of rectal bleeding and their attitudes towards seeking expert opinion for possible diagnostic testing for colorectal cancer (CRC)
Colonoscopy referral triggers among General Practitioners (GP) | 60 days
  To seeks to examine the GPs' perceived barriers to colonoscopy for patients with bleeding per rectum

IPD SHARING:
Plan to Share IPD: Undecided
Yes